CLINICAL TRIAL: NCT05234294
Title: Short and Long Term Symptoms After Omicron Infection in the Faroe Islands
Brief Title: Long Covid After COVID-19 Infection With Omicron Variant
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Faroese Hospital System (Other)
Collaborators: Chief Medical Officer's Office Faroe Islands (Unknown); University of the Faroe Islands (Other); National Hospital of the Faroe Islands (Other Government)
Responsible Party: Principal Investigator, Maria Skaalum Petersen, Phd, Faroese Hospital System
Other Study IDs: Omicron
Record Dates: First submitted 2022-02-09; First posted 2022-02-10 (Actual); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Omicron cases: All confirmed COVID-19 cases during January 2022 in the Faroe Islands
  Interventions: Other: Survey
- Controls: Participants in previous serological surveys during 2020 in the Faroe Islands.
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — We will investigate symptoms through monthly surveys.

SUMMARY:
The COVID-19 pandemic has led to a high disease burden worldwide, both during the acute disease phase and a large group of infected suffering from Long Covid. Long Covid has been subject to a lot of research, even though there is still much not understood. However, the need for time to pass before symptoms can be assessed limits research into Long Covid on a longer timescale.

The worldwide pandemic has shifted after the emergence of the Omicron variant. The number of confirmed COVID cases worldwide has risen to unprecedented levels. Yet, hospitalizations and death do not increase at the same level as with previous variants.

The observed shift in the pandemic with the increasing number of infections with the Omicron variant leads to the urgent question about Long Covid after Omicron infection. This rise has also taken place in the Faroe Islands, with many infections during December 2021 and January 2022. The majority of infections during January 2022 in the Faroe Islands are expected to be of the Omicron variant, presenting the opportunity to investigate symptoms after infection with the Omicron variant.

In this study, we will invite all infected with COVID-19 during January 2022 in the Faroe Islands to answer an online survey regarding symptoms. This survey will be sent out once a month for a total of six times, both focusing on acute symptoms and Long Covid symptoms.

Concurrently, we will send an online survey to Faroese inhabitants recruited in two separate random COVID-19 serological surveys during 2020, which will act as controls.

The knowledge gathered during this study will rapidly bring understanding to the urgent question of Long Covid after Omicron infections. We know that the Omicron variant leads to fewer hospitalizations and death than previous variants, yet the question of Long Covid is still unanswered, and needs rapid answers.

DETAILED DESCRIPTION:
Objectives Primary objective: To investigate Long Covid symptoms after Omicron infection through monthly surveys for six months, compared to controls not infected.

Secondary objective: To investigate acute symptoms during Omicron infection through the first survey shortly after the infection.

Methods All confirmed COVID-19 patients in January 2022 will receive an invitation to participate in an online survey.

We will send the online surveys in two separate bulks. The individuals with confirmed COVID-19 during the first half of January will receive the online survey first, at the same time as half of the controls. The rest of the COVID-19 cases will receive it during the first half of February, along with the rest of the control group.

Outcomes Self-reported symptoms through the online survey compared to the symptoms in the control group.

Hospitalization. Death.

Statistical analyses We will report the results as numbers and percentages. We will stratify analyses by age groups, gender, and previous immunity through infection or vaccination.

Population The target population is all infected Faroese COVID-19 patients during January 2022, when Omicron is expected to make up the majority of cases.

Controls will be participants in two separate serological surveys with randomly selected individuals that have not had COVID-19 during December 2021 and January 2022

Variables for COVID-19 cases

* Date of infection
* Previous COVID-19 infection, date
* Vaccination status and dates of vaccination
* Self-reported symptoms during the acute phase of the infection, pre-made list by research group, rated as none, mild, moderate, and severe.
* Option to write in other symptoms.
* Weight and height
* Self-reported severity of the disease course, rated as asymptomatic, mild, moderate, and severe.
* Time to resolution of acute symptoms
* Background information, including education level, current occupational status, smoking, co-morbidities, medicine use, and self-reported health.
* Date of hospitalization, length of hospitalization, date of ICU, length of ICU, date of death.

Variables for controls

* Previous COVID-19 infection, date
* Vaccination status and dates of vaccination
* Self-reported symptoms during the last week, pre-made list by research group, rated as none, mild, moderate, and severe.
* Option to write in other symptoms.
* Weight and height
* Self-reported severity of the disease course, rated as asymptomatic, mild, moderate, and severe.
* Time to resolution of acute symptoms
* Background information, including education level, current occupational status, smoking, co-morbidities, medicine use, and self-reported health.

Publication The results will be published in international scientific journals and press releases on www.health.fo.

Perspectives There is an urgent need to investigate Long Covid after an Omicron infection. This study can provide rapid answers to this question.

Strengths of this planned study include the possibility of performing a nationwide survey and the rapid reporting of both long-term and short-term symptoms.

Limitations include the possibility of a low participation rate.

ELIGIBILITY:
Inclusion Criteria Cases:

* Confirmed COVID-19 during January 2022 in the Faroe Islands.

Exclusion Criteria Cases:

* Not reachable

Inclusion Criteria Controls:

* Participant in serological survey amongst random sample of Faroese inhabitants in 2020

Exclusion Criteria Cases:

* Confirmed COVID-19 during December 2021 or January 2022

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The target population is all infected Faroese COVID-19 patients during January 2022, when Omicron is expected to make up the majority of cases.
  Controls will be participants in two separate serological surveys with randomly selected individuals that have not had COVID-19 during December 2021 and January 2022
Sampling Method: Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2022-01-31 (Actual); Primary Completion 2022-08-07 (Estimated); Study Completion 2022-08-07 (Estimated)

PRIMARY OUTCOMES:
Long Covid after Omicron | 6 months
  Symptoms gathered through survey

SECONDARY OUTCOMES:
Acute symptoms during Omicron infection | 1 month
  Symptoms gathered through survey

OTHER OUTCOMES:
Death | 6 months
  Any death, but seperately analyze deaths caused by COVID-19 and other reasons.
Hospitalization | 6 months
  Any hospitalization, but seperately analyze hospitalizations caused by COVID-19 and other reasons.

CONTACTS AND LOCATIONS:
Locations (1):
- The Faroses Hospital System, Tórshavn, Faroe Islands

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared in order to protect the right of the participating individuals.